CLINICAL TRIAL: NCT05435469
Title: Study on the Changes of Coping Strategies With Stressful Events and Mental Health Level Among Adolescents Before and After COVID-19 Pandemic.
Brief Title: The Changes of Coping With Stressful Events Among Adolescents Under the COVID-19 Pandemic.
Status: Completed | Type: Observational
Sponsor: Wei XIA, PhD (Other)
Responsible Party: Sponsor-Investigator, Wei XIA, PhD, Associate Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Other Study IDs: L2022SYSU-HL-044
Record Dates: First submitted 2022-06-25; First posted 2022-06-28 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Coping Behavior; Mental Health Issue
Keywords: adolescent; pandemic; coping behavior; mental health; stressful life event
MeSH Terms: conditions — Psychological Well-Being | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Questionnaires assessed adolescents: ① Teenagers aged 14-25. ② Chinese nationality, who has lived in China since the outbreak of the COVID-19 epidemic, and has experienced or is experiencing the epidemic and its normalization. ③ Have the normal cognitive ability, expression ability, and social participation ability.
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Participants will be asked to respond to the demographic information sheet, Adolescent Self-Rating Life Events Check List, Coping Inventory For Stressful Situations, Social Skills Rating System, brief-symptom-inventory, and Wong and Law EI Scale.

SUMMARY:
This study aims to describe the changes in coping strategies used by adolescents for stressful life events under the background of epidemic normalization; and explore the causes of coping strategy changes of stressful life events under the background of normalization of the epidemic situation among adolescents.

DETAILED DESCRIPTION:
Under the special background of normalization of the epidemic situation, this paper describes and discusses the subjective feelings, changes in coping strategies, and causes of adolescent stressful life events, and puts forward a coping mechanism model of stressful adolescent events, which reflects the psychological changes of adolescent groups in the era of the epidemic situation and provides the basis for subsequent intervention measures.

ELIGIBILITY:
Inclusion Criteria:

* Aged 14-25
* Chinese nationality, who has lived in China since the outbreak of the COVID-19 epidemic, and has experienced or is experiencing the epidemic and its normalization.
* Have the normal cognitive ability, expression ability, and social participation ability.

Exclusion Criteria:

* Be diagnosed with psychological or mental illness.
* Incapacitated or unable to provide informed consent.
* Patients with severe diseases.

Ages: 14 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: General adolescents
Sampling Method: Non-Probability Sample
Enrollment: 4300 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Coping strategies used after the pandemic | Baseline
  The Coping strategies used by the adolescents for the stressful life events after the COVID-19 pandemic will be measured by Coping Inventory For Stressful Situations with the 21-items.
Coping strategies used before the pandemic | Baseline
  The Coping strategies used by the adolescents for the stressful life events before the COVID-19 pandemic will be measured by Coping Inventory For Stressful Situations with the 21-items.
Mental health | Baseline
  The mental health level of the adolescents will be measured by brief-symptom-inventory with 53-items.
Emotional Intelligence status | Baseline
  The Emotional Intelligence status of the adolescents will be measured by Wong and Law EI Scale with 16-items.

SECONDARY OUTCOMES:
Stressful Life Events after pandemic | Baseline
  The Stressful Life Events experienced by the adolescents after the COVID-19 pandemic will be measured by Adolescent Self-Rating Life Events Check List with the 27-items.
Stressful Life Events before pandemic | Baseline
  The Stressful Life Events experienced by the adolescents before the COVID-19 pandemic will be measured by Adolescent Self-Rating Life Events Check List with the 27-items.
Social support | Baseline
  The social support that the adolescent could approach will be measured by Social Skills Rating System with the 10-items.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Xia, PhD, Principal Investigator — Sun Yat-sen University
Locations (1):
- XIAW, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
The non-identified IPD will be shared after the outcomes have been published.
Supporting Information: SAP
Time Frame: After the publication of the study
Access Criteria: Researchers should contact the PI for approval of the study protocol.

REFERENCES:
- [Derived] Ding H, Xu Z, Hu W, Guo Y, Wang C, Li S, Hui Z, Wang J, Peng X, Xia W. Changes of stressful life events, coping strategies and mental health among youths in the pre- and post-coronavirus 2019 pandemic era: A cross-sectional study. Int J Soc Psychiatry. 2023 Dec;69(8):2018-2030. doi: 10.1177/00207640231188321. Epub 2023 Aug 1. PMID 37528555